CLINICAL TRIAL: NCT03007667
Title: The Impact of Colorectal Cancer Surgery on Localization of Ureters; Prospective Clinical Trail
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ulas Aday, Director,Depertmant of Gastroenterological Surgery, Principal Investigator, Clinical M.D, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2016.4/2-13
Record Dates: First submitted 2016-12-30; First posted 2017-01-02 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: The Relocation of the Ureter After Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Colorectal cancer patients: Colorectal cancer patients

SUMMARY:
To investigate the changes in the anatomical location of ureters after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Curative surgery for colorectal cancer diagnosis

Exclusion Criteria:

1. Abnormal renal function
2. Not having the test in accordance with the cancer follow-up program
3. Contrast allergy
4. Any surgery for the ureters in history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08-15 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
relocation of ureters (milimeters) | 1/10/2016- 1/06/2017

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Koşuyolu Higher Specialization Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)